CLINICAL TRIAL: NCT03105479
Title: A Prospective, Multicenter Study to Investigate the Pharmacokinetics, Safety, and Efficacy of Cadazolid Versus Vancomycin in Pediatric Subjects With Clostridium Difficile-associated Diarrhea
Brief Title: Comparison of Cadazolid Versus Vancomycin in Children With Clostridium Difficile-associated Diarrhea (CDAD)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study suspended in October 2017 and terminated April 17, 2018 after decision to discontinue the study drug development
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC-061A303; 2015-004805-17 (EudraCT Number)
Record Dates: First submitted 2017-03-23; First posted 2017-04-10 (Actual); Results first posted 2019-04-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Clostridium Difficile Infection
Keywords: vancomycin; children; cadazolid; clostridium difficile associated diarrhea
MeSH Terms: conditions — Clostridium Infections | interventions — cadazolid; Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor masking in Part B only (no masking in Part A)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A / Cohort A (Experimental): Subjects from 12 years to 18 years old (exclusive) will receive cadazolid 500 mg per day for 10 days. The dose may be adjusted based on the pharmacokinetic (PK) and safety data reviewed for the first 3 subjects.
  Interventions: Drug: Cadazolid
- Part A / Cohort B (Experimental): Subjects from 6 years to 12 years old (exclusive) will receive cadazolid for 10 days. The dose will depend on the PK and safety data from cohort A reviewed by the Independent Data Monitoring Committee (IDMC).
  Interventions: Drug: Cadazolid
- Part A / Cohort C (Experimental): Subjects from 2 years to 6 years old (exclusive) will receive cadazolid for 10 days. The dose will depend on the PK and safety data from cohort B reviewed by the IDMC.
  Interventions: Drug: Cadazolid
- Part A/ Cohort D (Experimental): Subjects from 3 months to 2 years old (exclusive) will receive cadazolid for 10 days. The dose will depend on the PK and safety data from cohort C reviewed by the IDMC.
  Interventions: Drug: Cadazolid
- Part A/ Cohort E (Experimental): Subjects from birth to 3 months old (exclusive) will receive cadazolid for 10 days. The dose will depend on the PK and safety data from cohort D reviewed by the IDMC.
  Interventions: Drug: Cadazolid
- Part B / Cadazolid (Experimental): Subjects from birth to 18 years old (exclusive) will receive cadazolid for 10 days, at the dose defined in the corresponding age cohort in Part A.
  Interventions: Drug: Cadazolid
- Part B / Vancomycin (Active Comparator): Subjects from birth to 18 years old (exclusive) will receive vancomycin capsule (for subjects able to swallow) or vancomycin solution (for the others) during 10 days .
  Interventions: Drug: Vancomycin capsule; Drug: Vancomycin solution

INTERVENTIONS:
Drug: Cadazolid — Granules for oral suspension to be administered twice daily
  Other Names: ACT-179811
  Arms: Part A / Cohort A; Part A / Cohort B; Part A / Cohort C; Part A/ Cohort D; Part A/ Cohort E; Part B / Cadazolid
Drug: Vancomycin capsule — Capsule containing 125 mg of vancomycin to be administered orally 4 times a day
  Arms: Part B / Vancomycin
Drug: Vancomycin solution — Vancomycin powder to be administered as oral solution at a dose of 40 mg/kg/day, 3 to 4 times a day
  Arms: Part B / Vancomycin

SUMMARY:
Cadazolid has demonstrated activity against a bacteria named Clostridium difficile in animal studies. The results of a first study conducted in adult patients have suggested efficacy of the new antibiotic, cadazolid, in the treatment of diarrhea caused by this bacteria. This is the first study of cadazolid in children. The overall purpose of this study is to provide reassurance on the safety and efficacy of cadazolid in children suffering from infection due to Clostridium difficile.

DETAILED DESCRIPTION:
This multicenter, study will be run into two parts. Both parts will be run in consecutive age cohorts, starting from the oldest age categories(12 to < 18 years old) to the youngest (birth to < 3 months).

* Part A is an open-label, dose finding part to be conducted in at least 24 subjects.
* Part B follows a randomized, assessor-blinded, parallel-group design with vancomycin used as an active comparator. Part B will be conducted in about 176 children.

In both parts, the treatment period will be 10 days and will be followed by a Follow-up period of 28-32 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent by parents or legally authorized representatives (LAR) and assent by the child according to local requirements prior to initiation of any study-mandated procedure.
* Male or female from birth to < 18 years of age, diagnosed with Clostridium Difficile-associated diarrhea (CDAD).
* Females of childbearing potential must have a negative pregnancy test at screening and must agree to use an adequate and reliable method of contraception.

Key Exclusion Criteria:

* Positive Rotavirus test for subjects < 5 years.
* Fulminant or life-threatening CDAD.
* More than one previous episode of CDAD in the 3 month period prior to enrollment / randomization.
* Antimicrobial treatment active against CDAD administered within 24 h prior to screening except for metronidazole treatment failures (MTF).
* Subjects with body weight < 3 kg.
* Inflammatory bowel disease, chronic abdominal pain, or chronic diarrhea of any etiology.
* Fecal microbiota transplant (FMT), immunoglobulin therapy, or any investigational drug to prevent or treat CDAD within 1 month period (or 5 half-lives in case of investigational drug, whichever is longer) prior to enrollment / randomization.
* Monoclonal antibodies against C. difficile within 6 months prior to enrollment / randomization.
* Previous vaccination against C. difficile.
* Known mental disorders.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study, or compliance with the protocol.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (5):
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - University of Chicago, Dept. Of Medicine, Chicago, Illinois
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - SUNY Upstate Medical University - Upstate Golisano Children's Hospital (GCH) - Pediatric Designated AIDS Center, Syracuse, Ohio
  - Texas Children's Hospital Feigin Cente, Houston, Texas
- Universitair Ziekenhuis Brussel - Kinderziekenhuis, Jette, Belgium
- Infection Prevention & Control, AGW5 Foothills Medical Center 1403 29th Street N.W., Calgary, Canada
- FN Brno, Brno, Czechia
- Hungary (2):
  - Egyesített Szent István és Szent László Kórház - Rendelőintézet / Gyermekinfektológiai Osztály, Budapest
  - Pándy Kálmán Megyei Kórház, Gyula
- Italy (2):
  - Ospedale Buzzi, Milan
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale Pediatrico Bambino Gesu, Roma
- Poland (4):
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. Tadeusza Browicza, Bydgoszcz
  - Specjalistyczny Zespół Opieki Zdrowotnej nad Matką i Dzieckiem, Poznan
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Klinika Gastroenterologii, Hepatologii, Zaburzeń Odżywiania i Pediatrii, Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw
- Romania (2):
  - Institutul National De Boli Infectioase "Prof. Dr. Matei Bals", sectia IX pediatrie, Bucharest
  - Spitalul Clinic de Boli Infectioase "Sfanta Parascheva" Iasi, Clinica de Boli Infectioase I,, Iași
- Spain (2):
  - Hospital Sant Joan de Déu, Esplugues, Barcelona
  - Hospital Universitario Infantil LA PAZ, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to early termination of the study after sponsor's decision to discontinue the development of cadazolid, only one patient was enrolled at one site in the US.
Groups:
- Part A / Cohort A: Subjects from 12 years to 18 years old (exclusive) are to be treated with cadazolid 250 mg twice daily for 10 days. The dose may be adjusted based on the pharmacokinetic (PK) and safety data reviewed for the first 3 subjects.
- Part A / Cohort B: Subjects from 6 years to 12 years old (exclusive) are to be treated with cadazolid for 10 days (dose determined based on the PK and safety data from cohort A reviewed by the Independent Data Monitoring Committee (IDMC)).
- Part A / Cohort C: Subjects from 2 years to 6 years old (exclusive) are to be treated with cadazolid for 10 days. (dose determined based on the PK and safety data from cohort B reviewed by the IDMC).
- Part A/ Cohort D: Subjects from 3 months to 2 years old (exclusive) are to be treated with cadazolid for 10 days (dose determined based on the PK and safety data from cohort B reviewed by the IDMC).
- Part A/ Cohort E: Subjects from birth to 3 months old (exclusive) are to be treated with cadazolid for 10 days (dose determined based on the PK and safety data from cohort B reviewed by the IDMC). .
- Part B / Cadazolid: Subjects from birth to 18 years old (exclusive) are to be treated with cadazolid for 10 days, at the dose defined in the corresponding age cohort in Part A.
- Part B / Vancomycin: Subjects from birth to 18 years old (exclusive)are to be treated with vancomycin for 10 days either as capsules (for subjects able to swallow) or oral solution (for the others) .
Period: Overall Study
Arm/Group | Part A / Cohort A | Part A / Cohort B | Part A / Cohort C | Part A/ Cohort D | Part A/ Cohort E | Part B / Cadazolid | Part B / Vancomycin
Started | 1 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only one subject was enrolled in Part A. Part B was not conducted due to early study termination. Consequently the baseline characteristics are from one subject only.
Arm/Group | Part A / Cohort A
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12 years to < 18 years) | 1
  Children (2 years to < 12 years | 0
  infants and toddlers (3 months to < 2 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate During Part B
Description: This is the percentage of participants in part B reported as with a clinical cure. Clinical Cure is defined as: • <3 unformed bowel movement (UBM) per day (or no water diarrhea if subjects < 2 years of age), for at least 2 consecutive days between first dose of study treatment up to end of treatment (EOT) (inclusive) AND • Subject remains well up to EOT + 2 days (inclusive) based on investigator judgment AND • No need for additional antimicrobial treatment active against Clostridium difficile-associated diarrhea (CDAD) between first dose of study treatment up to EOT + 2 days (inclusive). percentage of subjects with a clinical cure
Time Frame: Day 10 (End of Treatment) + 2 days
Population: Due to the premature study termination, no subject was enrolled into Part B and consequently the percentage of subjects with a clinical cure could not be reported.
Groups:
- Part B: Due to early termination of the study, no subject was enrolled into Part B.
Arm/Group | Part B
Number analyzed (Participants) | 0

2. Primary Outcome: Maximal Plasma Concentration (Cmax) of Cadazolid During Part A
Description: Blood samples are collected at different timepoints on Day 10 for the determination of cadazolid Cmax after 10 days of treatment.
Time Frame: Day 10 (End of Treatment)
Population: Due to the premature study termination, cadazolid concentrations were obtained from only one subject and pharmacokineitc plasma profile was not analyzed because of lack of meaningful data.
Groups:
- Part A / Cohort A: One Subject aged between 12 and 18 years old received cadazolid 500 mg per day for 10 days.
Arm/Group | Part A / Cohort A
Number analyzed (Participants) | 0

3. Primary Outcome: Time to Reach Cmax (Tmax) of Cadazolid During Part A
Description: Blood samples are collected at different timepoints to determine the time when the maximal plasma concentration of cadazolid is reached.
Time Frame: Day 10 (End of Treatment)
Population: as for outcome 2
Arm/Group | Part A / Cohort A
Number analyzed (Participants) | 0

4. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) of Cadazolid During Part A
Description: Blood samples are collected at different timepoints for the determination of the cadazolid AUC over one dosing interval (0-12h) on Day 10.
Time Frame: Day 10 (End of Treatment)
Population: as for outcome 2
Arm/Group | Part A / Cohort A
Number analyzed (Participants) | 0

5. Primary Outcome: Fecal Concentrations of Cadazolid During Part A
Description: A fecal sample is collected as the end-of-treatment visit in all participants in Part A.
Time Frame: Day 10 (End of Treatment)
Population: Due to premature termination, fecal sample was collected from only one subject, consequently mean values cannot be provided and no statistical analyses can be performed.
Measure: Number; unit: mcg/g
Arm/Group | Part A / Cohort A
Number analyzed (Participants) | 1
mcg/g | 4520

6. Secondary Outcome: Clinical Cure Rate During Part A
Description: This is the percentage of participants in Part A reported as with a clinical cure. Clinical Cure is defined as: • <3 unformed bowel movement (UBM) per day (or no water diarrhea if subjects < 2 years of age), for at least 2 consecutive days between first dose of study treatment up to end of treatment (EOT) (inclusive) AND • Subject remains well up to EOT + 2 days (inclusive) based on investigator judgment AND • No need for additional antimicrobial treatment active against Clostridium difficile-associated diarrhea (CDAD) between first dose of study treatment up to EOT + 2 days (inclusive).
Time Frame: Day 10 (End of Treatment) + 2 days
Population: Due to premature termination, data were collected from only one subject, consequently percentage of participants with clinical cure cannot be calculated and no statistical analyses can be performed
Arm/Group | Part A / Cohort A
Number analyzed (Participants) | 0

7. Secondary Outcome: Sustained Clinical Cure Rate During Part A and Part B
Description: This is the percentage of participants in Parts A and B reported as with sustained clinical cure. Sustained clinical cure is defined as • Clinical Cure and no Recurrence until 30 days after the last study drug intake (end of study).
Time Frame: Day 40 (on average)
Population: Due to the premature termination of the study and consequent lack of meaningful data, no analyses were performed.
Groups:
- Part A / Cohorts A to E: Only one subject was included in cohort A; no subject was enrolled in the other cohorts due to early study termination.
- Part B / Cadazolid: No subject was enrolled in cohort B due to early study termination.
Arm/Group | Part A / Cohorts A to E | Part B / Cadazolid
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Recurrence Rate During Part A and Part B
Description: This is the percentage of participants in Parts A and B assessed as having a recurrence out of subjects meeting the criteria for Clinical Cure. Recurrence is defined as: • Clinical Cure AND New episode of diarrhea with ≥ 3 UBMs (or watery diarrhea if subject < 2 years) on any day between EOT + 3 days and end of study AND • Stool test showing positive C. difficile (as defined in Inclusion Criterion 4), AND •Antimicrobial treatment active against CDAD started between EOT + 3 days and end of study.
Time Frame: Day 40 (on average)
Population: Due to the premature termination of the study and consequent lack of meaningful data, no analyses were performed.
Arm/Group | Part A / Cohorts A to E | Part B / Cadazolid
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Recurrence in Part B
Description: This it the time (in days) elapsed between the last dose of study drug and the onset day of new episode of diarrhea reported as Kaplan-Meier estimates (KM estimates)
Time Frame: Day 40 (on average)
Population: Due to premature termination, no subject was enrolled in Part B. Consequently, no data can be reported during Part B
Arm/Group | Part B
Number analyzed (Participants) | 0

10. Secondary Outcome: Time to Resolution of Diarrhea in Part B
Description: This is the time (in days) elapsed between the first dose of study treatment and the resolution of diarrhea and reported as Kaplan-Meier estimates (KM estimates). The date of resolution of Diarrhea (ROD) is defined as the date of the first day of the 2 consecutive days on treatment with < 3 UBM (or no watery diarrhea for subjects < 2 years of age). Time to ROD is the time (in days) elapsed between the first dose of study treatment and the ROD
Time Frame: Day 10
Population: Due to premature termination, data were collected from only one subject, consequently KM estimates cannot be calculated and no statistical analyses can be performed
Arm/Group | Part B
Number analyzed (Participants) | 0

11. Secondary Outcome: Adverse Events Leading to Premature Discontinuation of Study Treatment
Description: Number of participants who prematurely discontinued the study treatment due to an adverse event
Time Frame: Up to Day 10
Population: Due to premature termination, no subject was enrolled in Part B. Consequently, no data can be reported during Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part A / Cohorts A to E | Part B / Cadazolid
Number analyzed (Participants) | 1 | 0
Participants | 0 |

12. Secondary Outcome: Marked Abnormalities in Clinical Laboratory Parameters
Description: Number of participants with any marked abnormalities in laboratory parameters up to 7 days after end of treatment
Time Frame: Day 17 (on average)
Population: Due to premature termination, no subject was enrolled in Part B. Consequently, no data can be reported during Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part A / Cohorts A to E | Part B / Cadazolid
Number analyzed (Participants) | 1 | 0
Participants | 0 |

13. Secondary Outcome: Marked Abnormalities in Vital Signs
Description: Number of subjects with any treatment-emergent abnormalities in vital signs (up to 7 days after end of treatment)
Time Frame: Day 17 (on average)
Population: Due to premature termination, no subject was enrolled in Part B. Consequently, no data can be reported during Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part A / Cohorts A to E | Part B / Cadazolid
Number analyzed (Participants) | 1 | 0
Participants | 0 |

14. Secondary Outcome: Treatment-emergent Adverse Events (TEAES)
Description: Number of subjects with any TEAEs. A TEAE is any adverse event temporally associated with the use of study treatment (from study treatment initiation until 7 days after study treatment discontinuation) whether or not considered by the investigator as related to study treatment.
Time Frame: Day 17 (on average)
Population: Due to premature termination, no subject was enrolled in Part B. Consequently, no data can be reported during Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part A / Cohorts A to E | Part B / Cadazolid
Number analyzed (Participants) | 1 | 0
Participants | 0 |

ADVERSE EVENTS:
Time Frame: From study treatment initiation up to Day 37 (i.e., 27 days after the end of treatment)
Description: All adverse events (AE) which occurred at any time during the treatment period (10 days with cadazolid) and during the follow-up period (about 30 days) are reported. All AEs reported below occurred during the follow-up period.
Groups:
- Overall Study (Part A and Part B): Only one subject was included in cohort A; no subject was enrolled in the other cohorts of Part A or Part B due to early study termination.
Arm/Group | Overall Study (Part A and Part B)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (Part A and Part B) (N=1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only one subject was enrolled due to early study termination. Consequently results are not meaningful and no statistical analyses could be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation. Upon review, Actelion may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights.

DOCUMENTS (1):
  • Study Protocol (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT03105479/Prot_000.pdf